CLINICAL TRIAL: NCT00182143
Title: PROphylaxis for ThromboEmbolism in Critical Care Trial (PROTECT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Critical Care Trials Group (Other); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network)
Responsible Party: McMaster University, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ISRCTN54618366
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2007-10

CONDITIONS: Critical Illness; Deep Venous Thrombosis
Keywords: Critically Ill; Deep Venous ThromboEmbolism; Randomized Controlled Trial
MeSH Terms: conditions — Critical Illness; Venous Thrombosis | interventions — Heparin, Low-Molecular-Weight; Dalteparin; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMWH (Fragmin, dalteparin) (Active Comparator): Placebo dose (normal saline) = AM dose LMWH (Fragmin, dalteparin) 5000IU daily = PM dose
  Interventions: Drug: LMWH (Fragmin, dalteparin)
- 2 (Active Comparator): Unfractionated Heparin 5000IU BID
  Interventions: Drug: Unfractionated Heparin

INTERVENTIONS:
Drug: LMWH (Fragmin, dalteparin) — Placebo AM dose (normal saline) and LMWH (Fragmin, dalteparin) 5000IU PM dose
  Other Names: Fragmin
  Arms: LMWH (Fragmin, dalteparin)
Drug: Unfractionated Heparin — 5000 IU BID
  Other Names: Heparin Sodium
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of Low Molecular Weight Heparin (LMWH) (Fragmin, dalteparin) versus Unfractionated Heparin (UFH) on the primary outcome of proximal leg Deep Vein Thrombosis (DVT) diagnosed by compression ultrasound, and the secondary outcomes of Pulmonary Embolism (PE), bleeding, Heparin-Induced Thrombocytopenia (HIT), and objectively confirmed venous thrombosis at any site.

DETAILED DESCRIPTION:
PROTECT: The PROphylaxis for ThromboEmbolism in Critical Care Trial.

Background: Critically ill patients have an increased risk of deep venous thrombosis (DVT) due to their acute illness, procedures such as central venous catheterization, and immobility. Among patients in the intensive care unit (ICU), DVT is an important problem, since thrombus propagation and embolization can lead to potentially fatal pulmonary embolism (PE). Only 1 randomized trial (n=119) in medical-surgical ICU patients demonstrates that unfractionated heparin (UFH) prevents DVT compared to no prophylaxis; only 1 randomized trial (n=223) in ventilated COPD patients shows that low molecular weight heparin (LMWH) prevents DVT compared to no prophylaxis. In medical-surgical ICUs, the effect of LMWH vs UFH for DVT prevention has not been tested. On one hand, LMWH is likely to be more effective at venous thromboembolism (VTE) prevention and is associated with a lower rate of heparin-induced thrombocytopenia (HIT). On the other hand, UFH is likely associated with less bleeding, and is less expensive. Current guidelines indicate that in the absence of comparative data, both LMWH and UFH are suitable for thromboprophylaxis in this population, but that a randomized trial is needed.

PROTECT Pilot: In our Pilot Study, feasibility objectives were to assess:

1) timely enrolment and complete, blinded study drug administration, 2) the bioaccumulation of LMWH in patients with acquired renal insufficiency, 3) twice weekly leg ultrasounds, and 4) recruitment rates.

1. Timely, complete administration occurred for 98% of scheduled doses; every dose was blinded.
2. No LWMH bioaccumulation was observed.
3. Scheduled ultrasounds occurred without exception.
4. Recruitment will be 4 patients/month/centre after modification of 3 exclusion criteria in the PROTECT pilot.

Objective: To evaluate the effect of LMWH (dalteparin) vs UFH on the primary outcome of proximal leg DVT diagnosed by compression ultrasound, and the secondary outcomes of PE, bleeding, HIT, and objectively confirmed venous thrombosis at any site.

Design: Prospective randomized stratified concealed blinded multicentre trial.

Population: Inclusion Criteria: Eligible patients in medical-surgical ICUs will be >18 years old, weigh > 45 kg, and have an expected ICU stay > 72 hours.

Exclusion Criteria: Patients admitted to ICU post trauma, orthopedic surgery, or neurosurgery, with severe hypertension, DVT, PE or major hemorrhage within 3 months, International Normalized Ratio (INR) > 2 ULN, Partial Thromboplastin Time (PTT) > 2 ULN, platelets < 75 x 109/L, or those requiring therapeutic anticoagulation will be excluded. Patients with a contraindication to heparin, blood products or pork products, with > 3 days of LMWH or UFH in ICU, patients who are pregnant, undergoing withdrawal of life support, or are enrolled in this or a related trial will also be excluded.

Methods: Using centralized telephone randomization, we will allocate 3,650 patients in 40 centres to LMWH (dalteparin) 5,000 IU daily or UFH 5,000 IU twice daily SC for the duration of ICU stay. Patients, families, all clinicians and researcher will be blinded; only the pharmacist will be aware of allocation. Bilateral proximal leg compression ultrasounds will be performed within 48h of ICU admission, twice weekly, and on suspicion of DVT. PE will be diagnosed by a predefined diagnostic algorithm. We will record bleeding, HIT, other venous thrombosis and complications. Protocol adherence will be maximized using training, manuals, study aids, site visits, audit and feedback. Blinded Adjudication Committees will adjudicate endpoints. PROTECT will be conducted by the Canadian Critical Care Trials Group and overseen by an independent DSMB.

Relevance: The results of PROTECT will be used to develop evidence based practice guidelines regarding the safety and efficacy of LMWH (dalteparin) vs UFH for thromboprophylaxis in medical-surgical ICU patients around the world.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >/= 18 years of age
2. Actual body weight is >/= 45 kg
3. Admission to ICU expected to be >/= 72 hours in duration

Exclusion Criteria:

1. Neurosurgery within last 3 months
2. Ischemic stroke within last 3 months
3. Intracranial hemorrhage within last 3 months
4. Systolic Blood Pressure >/= 180mm Hg, Diastolic Blood Pressure >/= 110mm Hg for >/= 12 hours requiring vasoactive drug infusion
5. Major hemorrhage within last week unless definitively treated
6. Coagulopathy as defined by INR >/= 2 times upper limit of normal [ULN], or PTT >/= 2 times ULN, at time of screening
7. Thrombocytopenia defined as platelet count </= 75 x 109/L, at time of screening
8. Other heparin contraindications (e.g., HIT, pregnancy, lactating)
9. Contraindication to blood products (e.g., Jehovah's Witness)
10. Unable to perform lower limb ultrasound (e.g., bilateral above the knee amputation, or severe distal extremity burns)
11. Limitation of life support, Life expectancy </= 14 days, or palliative care
12. Contamination (e.g., >/= 3 doses of LMWH during this ICU admission)
13. Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3659 (Actual)
Dates: Start 2006-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of LMWH (Fragmin, dalteparin) versus UFH on the primary outcome of proximal leg DVT diagnosed by compression ultrasound | While in ICU to a maximum of 90 days

SECONDARY OUTCOMES:
To evaluate the effect of LMWH (Fragmin, dalteparin) versus UFH on the secondary outcomes of PE, bleeding, HIT, and objectively confirmed venous thrombosis at any site | While in ICU to a maximum of 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Cook, MD, Principal Investigator — McMaster University
Locations (67):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson, Houston, Texas
- Australia (17):
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Flinders Hospital, Bedford Park, Victoria
  - Bendigo Health Care, Bendigo, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Center, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Frankston Hospital, Frankston, Victoria
  - The Geelong Hospital, Geelong, Victoria
  - Austin Hill Hospital, Heidelburg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal North Shore Hospital, St Leonards
- Brazil (5):
  - UTI da Enfermaria de Clinical Medica do Hospital, São Paulo, Brazil
  - Hospitalar Santa Casa, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rs Cep
  - Hospital ProCardiaco, Rio de Janeiro
  - Hospital Coracao, São Paulo
- Canada (35):
  - Foothills Hospital, Calgary, Alberta
  - The Peter Lougheed Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Surry Memorial, Surrey, British Columbia
  - Royal Columbian Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health, Halifax, Nova Scotia
  - Guelph General Hospital, Guelph, Ontario
  - Hamilton Health Science Centre - Hamilton General Hospital, Hamilton, Ontario
  - Hamilton Health Science Centre - McMaster University, Hamilton, Ontario
  - St Joseph's HealthCare, Hamilton, Ontario
  - Hamilton Health Science Center - Henderson Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - London Health Science Center, London, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Ottawa Hospital - General Hospital, Ottawa, Ontario
  - Ottawa Hospital - Civic Site, Ottawa, Ontario
  - Sunnybrook and Women's College Health Science Centre, Toronto, Ontario
  - St Michaels Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Royal Victoria Hospital, McGill University Health Center, Montreal, Quebec
  - Montreal General Hospital, McGill University Health Centre, Montreal, Quebec
  - Hopital Sacre Couer, Montreal, Quebec
  - Hopital Charles LeMoyne, Montreal, Quebec
  - Hopital Maisonneuve, Montreal, Quebec
  - Centre Hospitalier Affilie-Enfant Jesus, Québec, Quebec
  - Hopital Laval, Québec, Quebec
  - Sherbrooke University (CHUS) Hospital, Sherbrooke, Quebec
- Saudi Arabia (5):
  - King Abdulaziz Medical City Hospital, Riyadh, Riyahd
  - King Abdulaziz University Hospital, Jeddah
  - King Faisal Specialist & Research Center, Jeddah
  - King Fahad Medical City, Riyadh
  - Riyadh Military Hospital, Riyadh
- Guys and St Thomas Hospital, London, England, United Kingdom

REFERENCES:
- [Derived] Li G, Cook DJ, Thabane L, Friedrich JO, Crozier TM, Muscedere J, Granton J, Mehta S, Reynolds SC, Lopes RD, Lauzier F, Freitag AP, Levine MA; PROTECT Investigators for the Canadian Critical Care Trials Group, and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Risk factors for mortality in patients admitted to intensive care units with pneumonia. Respir Res. 2016 Jul 11;17(1):80. doi: 10.1186/s12931-016-0397-5. PMID 27401184
- [Derived] Li G, Thabane L, Cook DJ, Lopes RD, Marshall JC, Guyatt G, Holbrook A, Akhtar-Danesh N, Fowler RA, Adhikari NKJ, Taylor R, Arabi YM, Chittock D, Dodek P, Freitag AP, Walter SD, Heels-Ansdell D, Levine MAH. Risk factors for and prediction of mortality in critically ill medical-surgical patients receiving heparin thromboprophylaxis. Ann Intensive Care. 2016 Dec;6(1):18. doi: 10.1186/s13613-016-0116-x. Epub 2016 Feb 27. PMID 26921148
- [Derived] Li G, Cook DJ, Levine MAH, Guyatt G, Crowther M, Heels-Ansdell D, Holbrook A, Lamontagne F, Walter SD, Ferguson ND, Finfer S, Arabi YM, Bellomo R, Cooper DJ, Thabane L; PROTECT Investigators for the Canadian Critical Care Trials Group, and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Competing Risk Analysis for Evaluation of Dalteparin Versus Unfractionated Heparin for Venous Thromboembolism in Medical-Surgical Critically Ill Patients. Medicine (Baltimore). 2015 Sep;94(36):e1479. doi: 10.1097/MD.0000000000001479. PMID 26356708
- [Derived] Fowler RA, Mittmann N, Geerts WH, Heels-Ansdell D, Gould MK, Guyatt G, Krahn M, Finfer S, Pinto R, Chan B, Ormanidhi O, Arabi Y, Qushmaq I, Rocha MG, Dodek P, McIntyre L, Hall R, Ferguson ND, Mehta S, Marshall JC, Doig CJ, Muscedere J, Jacka MJ, Klinger JR, Vlahakis N, Orford N, Seppelt I, Skrobik YK, Sud S, Cade JF, Cooper J, Cook D; Canadian Critical Care Trials Group; Australia and New Zealand Intensive Care Society Clinical Trials Group. Economic evaluation of the prophylaxis for thromboembolism in critical care trial (E-PROTECT): study protocol for a randomized controlled trial. Trials. 2014 Dec 20;15:502. doi: 10.1186/1745-6215-15-502. PMID 25528663
- [Derived] Crowther M, Cook D, Guyatt G, Zytaruk N, McDonald E, Williamson D, Albert M, Dodek P, Finfer S, Vallance S, Heels-Ansdell D, McIntyre L, Mehta S, Lamontagne F, Muscedere J, Jacka M, Lesur O, Kutsiogiannis J, Friedrich J, Klinger JR, Qushmaq I, Burry L, Khwaja K, Sheppard JA, Warkentin TE; PROTECT collaborators; Canadian Critical Care Trials Group; Australian and New Zealand Intensive Care Society Clinical Trials Group. Heparin-induced thrombocytopenia in the critically ill: interpreting the 4Ts test in a randomized trial. J Crit Care. 2014 Jun;29(3):470.e7-15. doi: 10.1016/j.jcrc.2014.02.004. Epub 2014 Feb 14. PMID 24726205
- [Derived] Lamontagne F, McIntyre L, Dodek P, Heels-Ansdell D, Meade M, Pemberton J, Skrobik Y, Seppelt I, Vlahakis NE, Muscedere J, Reece G, Ostermann M, Padayachee S, Alhashemi J, Walsh M, Lewis B, Schiff D, Moody A, Zytaruk N, Leblanc M, Cook DJ; Prophylaxis for Thromboembolism in Critical Care Trial Investigators; Canadian Critical Care Trials Group; Australian and New Zealand Intensive Care Society Clinical Trials Group. Nonleg venous thrombosis in critically ill adults: a nested prospective cohort study. JAMA Intern Med. 2014 May;174(5):689-96. doi: 10.1001/jamainternmed.2014.169. PMID 24638843
- [Derived] Lauzier F, Arnold DM, Rabbat C, Heels-Ansdell D, Zarychanski R, Dodek P, Ashley BJ, Albert M, Khwaja K, Ostermann M, Skrobik Y, Fowler R, McIntyre L, Nates JL, Karachi T, Lopes RD, Zytaruk N, Finfer S, Crowther M, Cook D. Risk factors and impact of major bleeding in critically ill patients receiving heparin thromboprophylaxis. Intensive Care Med. 2013 Dec;39(12):2135-43. doi: 10.1007/s00134-013-3044-3. Epub 2013 Aug 14. PMID 23942857
- [Derived] Smith OM, McDonald E, Zytaruk N, Foster D, Matte A, Clarke F, Fleury S, Krause K, McArdle T, Skrobik Y, Cook DJ. Enhancing the informed consent process for critical care research: strategies from a thromboprophylaxis trial. Intensive Crit Care Nurs. 2013 Dec;29(6):300-9. doi: 10.1016/j.iccn.2013.04.006. Epub 2013 Jul 18. PMID 23871290
- [Derived] Williamson DR, Albert M, Heels-Ansdell D, Arnold DM, Lauzier F, Zarychanski R, Crowther M, Warkentin TE, Dodek P, Cade J, Lesur O, Lim W, Fowler R, Lamontagne F, Langevin S, Freitag A, Muscedere J, Friedrich JO, Geerts W, Burry L, Alhashemi J, Cook D; PROTECT collaborators, the Canadian Critical Care Trials Group, and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Thrombocytopenia in critically ill patients receiving thromboprophylaxis: frequency, risk factors, and outcomes. Chest. 2013 Oct;144(4):1207-1215. doi: 10.1378/chest.13-0121. PMID 23788287
- [Derived] Smith OM, McDonald E, Zytaruk N, Foster D, Matte A, Clarke F, Meade L, O'Callaghan N, Vallance S, Galt P, Rajbhandari D, Rocha M, Mehta S, Ferguson ND, Hall R, Fowler R, Burns K, Qushmaq I, Ostermann M, Heels-Ansdell D, Cook D; PROTECT Research Coordinators; PROTECT Investigators; Canadian Critical Care Trials Group; Australian, New Zealand Intensive Care Society Clinical Trials Group. Rates and determinants of informed consent: a case study of an international thromboprophylaxis trial. J Crit Care. 2013 Feb;28(1):28-39. doi: 10.1016/j.jcrc.2012.08.005. Epub 2012 Oct 22. PMID 23089679
- [Derived] Cook D, Meade M, Guyatt G, Walter SD, Heels-Ansdell D, Geerts W, Warkentin TE, Cooper DJ, Zytaruk N, Vallance S, Berwanger O, Rocha M, Qushmaq I, Crowther M. PROphylaxis for ThromboEmbolism in Critical Care Trial protocol and analysis plan. J Crit Care. 2011 Apr;26(2):223.e1-9. doi: 10.1016/j.jcrc.2011.02.010. PMID 21482348
- [Derived] PROTECT Investigators for the Canadian Critical Care Trials Group and the Australian and New Zealand Intensive Care Society Clinical Trials Group; Cook D, Meade M, Guyatt G, Walter S, Heels-Ansdell D, Warkentin TE, Zytaruk N, Crowther M, Geerts W, Cooper DJ, Vallance S, Qushmaq I, Rocha M, Berwanger O, Vlahakis NE. Dalteparin versus unfractionated heparin in critically ill patients. N Engl J Med. 2011 Apr 7;364(14):1305-14. doi: 10.1056/NEJMoa1014475. Epub 2011 Mar 22. PMID 21417952
- See also: PROTECT Collaborator Web Page — http://clarityresearch.ca/protect/protect_trial/